CLINICAL TRIAL: NCT01256450
Title: A 12-Week, Placebo Controlled, Double Blind, Randomized Withdrawal Study to Evaluate the Efficacy and Safety of Buprenorphine HCl Buccal Film in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety Study of Buprenorphine HCl Buccal Film in Subjects With Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUP-301
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Pain; Low Back Pain
Keywords: buccal soluble film; enriched enrollment; randomized withdrawal
MeSH Terms: conditions — Pain; Low Back Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BEMA Buprenorphine (Experimental): buprenorphine buccal soluble film
  Interventions: Drug: Buprenorphine
- BEMA Placebo (Placebo Comparator): placebo buccal soluble film
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — buccal soluble film; applied to the buccal mucosa twice daily
  Other Names: buprenorphine buccal soluble film; BEMA Buprenorphine; BELBUCA; buprenorphine HCl buccal film
  Arms: BEMA Buprenorphine
Drug: Placebo — buccal soluble film; applied to the buccal mucosa twice daily
  Other Names: Placebo buccal soluble film; Placebo buccal film; BEMA placebo
  Arms: BEMA Placebo

SUMMARY:
The purpose of this study is to determine whether buprenorphine hydrochloride (HCl) buccal film is effective and safe in the treatment of chronic low back pain (CLBP).

DETAILED DESCRIPTION:
This is an enriched enrollment, randomized withdrawal study with an open label, dose-titration period followed by a randomized, double-blind, placebo-controlled treatment period of 12 weeks. During the double-blind treatment period, this study will evaluate the effectiveness of buprenorphine HCl buccal film versus placebo buccal film in treating CLBP in subjects.

Buprenorphine HCl buccal film is an oral transmucosal form of the opioid analgesic, buprenorphine hydrochloride, intended for application to the buccal mucosa. Buprenorphine is a synthetic opioid that is classified as a partial µ-receptor agonist and a Schedule III controlled substance in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-nursing female aged 18 or older
* History of moderate to severe chronic low back pain for ≥3 months with a pain intensity ≥5 [11 point numerical rating scale] reported at the open-label titration period Day 0/1 visit following a washout period (opioids, nonsteroidal anti-inflammatory drugs [NSAIDs], and muscle relaxants) of approximately 12 to 24 hours
* Currently taking ≤60 mg oral morphine/day or equianalgesic dose of another opioid (including opioid naïve) for 1 week or longer
* Stable health, as determined by the Investigator, on the basis of medical history, physical examination, and screening laboratory results so as to comply with all study procedures
* Female subjects of childbearing potential must be using a recognized effective method of birth control
* Written informed consent obtained at Screening, prior to any procedure being performed

Exclusion Criteria:

* Reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, meningitis, and discitis
* Surgical procedure for back pain within 2 months prior to screening or nerve/plexus block within 4 weeks of screening
* Hypokalemia or clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia
* Corrected QT (QTc) interval of >450 milliseconds on the 12-lead electrocardiogram (ECG)
* History of long QT syndrome, or an immediate family member with this condition
* Diagnosis of moderate to severe hepatic impairment.
* History of severe emesis with opioids
* Clinically significant sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Finn, PharmD, Study Director — BioDelivery Sciences International, Inc.
Locations (24):
- United States (24):
  - Alabama Orthopaedic Center - Research, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - University of California, San Diego Medical Center, UCSD Center for Pain Medicine, La Jolla, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Taylor Research, LLC, Marietta, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - International Clinical Research Institute, Leawood, Kansas
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - Research Across American, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Allegheny Pain Management, Altoona, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Southwest Urgent Care Center, El Paso, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 334 subjects who were enrolled in the open-label (OL) titration phase; a total of 235 completed the open-label titration phase and were randomized in the double-blind (DB) treatment phase.
Groups:
- OL Buprenorphine HCl Buccal Film: Buprenorphine hydrochloride (HCl) buccal film, 60, 120, 180, or 240 µg, applied to the buccal mucosa every 12 hours for up to 4 weeks in the open-label titration period
- DB Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 60, 120, 180, or 240 µg, applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment period
- DB Placebo Film: Placebo buccal film applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind treatment period
Period: Open-label Titration
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Started | 334 | 0 | 0
Completed | 235 | 0 | 0
Not Completed | 99 | 0 | 0
Not completed — Adverse Event | 39 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0
Not completed — Lack of analgesic effect | 30 | 0 | 0
Not completed — Non-compliance | 9 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0
Not completed — Other | 13 | 0 | 0
Period: Double-blind Treatment
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Started | 0 (All subjects completing OL titration in the previous period were randomized to a DB treatment.) | 117 (Subjects were randomized to DB treatment after completing OL titration in the previous period.) | 118 (Subjects were randomized to DB treatment after completing OL titration in the previous period.)
Completed | 0 | 89 | 81
Not Completed | 0 | 28 | 37
Not completed — Adverse Event | 0 | 8 | 6
Not completed — Lost to Follow-up | 0 | 1 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lack of analgesic effect | 0 | 5 | 6
Not completed — Non-compliance | 0 | 5 | 4
Not completed — Opioid withdrawal symptoms | 0 | 0 | 1
Not completed — Other | 0 | 9 | 12

BASELINE CHARACTERISTICS:
Population: Analysis based on Randomized population; all subjects who were randomized into the double-blind period, even if study drug was not taken in the period
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film | Total
Number analyzed (Participants) | 117 | 118 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 17 | 18 | 35
Age, Continuous [Median (Full Range); unit: years] | 52.0 [21 to 89] | 51.5 [20 to 77] | 52.0 [20 to 89]
Gender [Count of Participants; unit: Participants]
  Female | 62 | 66 | 128
  Male | 55 | 52 | 107
Region of Enrollment [Number; unit: participants]
  United States | 117 | 118 | 235

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity From Baseline to Week 12
Description: Change in pain intensity = average of daily pain scores from the last 7 days prior to week 12 visit - average of daily pain scores for the last 7 days prior to randomization. Average pain intensity over the last 24 hours was rated on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Baseline, Week 12
Population: Analysis based on Intent-to-Treat (ITT) population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale | 0.33 (1.944) | 0.46 (2.093)
Statistical Analysis 1: Comparison: DB Buprenorphine HCl Buccal Film vs DB Placebo Film; Test type: Superiority or Other; p = .5870, ANCOVA; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.646 to 0.366]

2. Secondary Outcome: Change From Baseline in Pain Intensity Over Time Using NRS Scale
Description: Change in pain intensity = average of daily pain scores from the last 7 days prior to each visit - average of daily pain scores for the last 7 days prior to randomization. Average pain intensity over the last 24 hours was rated on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Baseline; Day 14, Day 28, Day 42, Day 56, Day 70, and Day 84
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale
  Day 14 | 0.21 (1.469) | 0.25 (1.624)
  Day 28 | 0.20 (1.539) | 0.29 (1.877)
  Day 42 | 0.13 (1.535) | 0.25 (1.840)
  Day 56 | 0.21 (1.709) | 0.23 (1.926)
  Day 70 | 0.15 (1.783) | 0.35 (2.056)
  Day 84 | 0.29 (1.984) | 0.38 (2.058)

3. Secondary Outcome: Number of Participants With Response to Treatment as Assessed by an NRS Scale
Description: Responses are defined as the relative improvement in pain score at week 12 from baseline, calculated from ratings of average pain intensity over the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Number; unit: participants
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
participants
  ≥0% Response | 117 | 118
  ≥10% Response | 48 | 32
  ≥20% Response | 37 | 30
  ≥30% Response | 28 | 27
  ≥40% Response | 19 | 23
  ≥50% Response | 13 | 20
  ≥60% Response | 11 | 16
  ≥70% Response | 8 | 13
  ≥80% Response | 5 | 9
  ≥90% Response | 5 | 7
  ≥100% Response | 3 | 6

4. Secondary Outcome: Percentage of Participants With Treatment Failure in the Double-blind Treatment Phase (up to 12 Weeks)
Description: Treatment failure is defined as study discontinuation due to lack of efficacy or due to adverse event in the double-blind treatment phase.
Time Frame: Baseline to treatment failure or end of double-blind treatment phase (up to 12 weeks)
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
percentage of participants | 9.4 | 11.9

5. Secondary Outcome: Subject Impression of Change in Pain Intensity From Baseline to Week 12 Using PGIC Scale
Description: Subjects assessed changes in activity, limitations, symptoms, and overall quality of life related to their painful condition since beginning treatment using the Patient Global Impression of Change (PGIC), a balanced 7-point scale from 1 (no change or condition got worse) to 7 (a great deal better and considerable improvement that has made all the difference).
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale | -0.32 (2.091) | -0.92 (2.110)

6. Secondary Outcome: Change From Baseline to Week 12 in Treatment Satisfaction Using TSQM
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) is a 14-item instrument used to assess the subject's satisfaction with the ability of the study medication to prevent or treat the condition of chronic low back pain (CLBP) for effectiveness, side effects, convenience, and global satisfaction. Scores range from 0 to 100, where a higher score indicates less dissatisfaction (ie, greater satisfaction).
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale
  Effectiveness | -2.06 (25.172) | -9.03 (27.804)
  Side effects | 3.09 (14.137) | 10.88 (18.243)
  Convenience | -3.12 (13.294) | -0.00 (14.081)
  Global satisfaction | -8.19 (26.146) | -11.73 (26.829)

7. Secondary Outcome: Change From Baseline to Week 12 in Roland Morris Disability Questionnaire
Description: Subjects assess disability due to back pain using the Roland Morris Disability Questionnaire (RMDQ) consisting of 24 statements of disability. The score of the RMDQ is the total number of items checked, ranging from 0 to 24 with higher scores indicating greater disability.
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale | 0.09 (5.606) | 1.00 (4.319)

8. Secondary Outcome: Change From Baseline to Week 12 in Subject's Overall Satisfaction With Study Drug
Description: Subjects were asked to rate their overall satisfaction with their study drug on a 5-point scale ranging from 1 (poor) to 5 (excellent).
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale | -0.30 (1.409) | -0.48 (1.329)

9. Secondary Outcome: Change From Baseline to Week 12 in Investigator's Overall Satisfaction With Study Drug
Description: Investigators rated their overall satisfaction with the study drug administered to a given subject on a 5-point scale ranging from 1 (poor) to 5 (excellent).
Time Frame: Baseline, Week 12
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
units on a scale | -0.27 (1.312) | -0.37 (1.369)

10. Secondary Outcome: Use of Rescue Medication
Description: Calculated from the use of rescue medication recorded in subject diary as the sum of all rescue medication tablets used in the last 7 days previous to the derived visit, divided by the number of days in this duration where the amount was reported.
Time Frame: Day 7, 14, 28, 42, 56, 70, 84, and 91 within double-blind treatment phase
Population: Analysis based on ITT population; all randomized subjects who received at least 1 dose of double-blind study medication
Measure: Mean (Standard Deviation); unit: Tablets per day
Arm/Group | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Number analyzed (Participants) | 117 | 118
Tablets per day
  Day 7 | 0.87 (1.143) | 0.82 (1.103)
  Day 14 | 0.93 (1.135) | 1.03 (1.289)
  Day 28 | 0.93 (1.239) | 1.02 (1.325)
  Day 42 | 0.97 (1.250) | 1.04 (1.358)
  Day 56 | 0.89 (1.245) | 0.99 (1.364)
  Day 70 | 0.83 (1.197) | 0.98 (1.611)
  Day 84 | 0.97 (1.277) | 0.91 (1.276)
  Follow-up Day 91 | 0.79 (1.143) | 1.07 (1.370)

ADVERSE EVENTS:
Time Frame: From study drug dispensing in open-label titration phase to about 1 week after last dose (Day 91/follow-up visit) in the double-blind phase, up to 17 weeks
Description: Analysis for open-label titration phase based on Safety population; all enrolled subjects who receive at least 1 dose of study drug. Analysis for double-blind treatment phase is based on Randomized population; all subjects who were randomized into double-blind treatment, even if study drug was not taken.
Groups:
- OL Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 60, 120, 180, or 240 µg, applied to the buccal mucosa every 12 hours for up to 4 weeks in the open-label titration period
- DB Buprenorphine HCl Buccal Film: Buprenorphine HCl buccal film, 60, 120, 180, or 240 µg, applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind period
- DB Placebo Film: Placebo buccal film applied to the buccal mucosa every 12 hours for 12 weeks in the double-blind period
Arm/Group | OL Buprenorphine HCl Buccal Film | DB Buprenorphine HCl Buccal Film | DB Placebo Film
Serious Adverse Events (participants affected / at risk) | 1/330 | 1/117 | 0/118
Other Adverse Events (participants affected / at risk) | 163/330 | 36/117 | 28/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL Buprenorphine HCl Buccal Film (N=330) | DB Buprenorphine HCl Buccal Film (N=117) | DB Placebo Film (N=118)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL Buprenorphine HCl Buccal Film (N=330) | DB Buprenorphine HCl Buccal Film (N=117) | DB Placebo Film (N=118)
CONSTIPATION (Gastrointestinal disorders) | 36 (37) | 7 (7) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 108 (118) | 11 (11) | 10 (11)
VOMITING (Gastrointestinal disorders) | 19 (19) | 6 (7) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 7 (7) | 3 (3) | 7 (7)
DIZZINESS (Nervous system disorders) | 30 (35) | 4 (4) | 1 (1)
HEADACHE (Nervous system disorders) | 39 (45) | 12 (14) | 5 (6)
INSOMNIA (Psychiatric disorders) | 8 (9) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The oral or written use of study results by the Investigator is not permitted without the express written consent from the Sponsor.